CLINICAL TRIAL: NCT02424279
Title: Invasive Treatment of Pain Associated With Pancreatic Cancer on Different Levels of WHO Analgesic Ladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Łukasz Dobosz, MD, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUG10
Record Dates: First submitted 2015-01-02; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Cancer; Pain
Keywords: pancreatic cancer; pain; splanchnicectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical treatment (Active Comparator): Patients from the first group will undergo thoracoscopic splanchnicectomy. The surgery will be performed in general anaesthesia, with tracheal intubation in prone position. The greater splanchnic nerve will be identified at its origin in sympathetic trunk, dissected together with all collaterals all the way down to the diaphragm and excised. Additional splanchnic nerves (smaller, minimus) will be incised or excised if connected to the greater splanchnic nerve. Single sutures will be applied to the skin. Then the procedure will be repeated on the contralateral side.
  Interventions: Procedure: Splanchnicectomy
- Conservative Treatment (No Intervention): Patients from the second group will be offered best available conservative pain treatment. The list of medication on stage 1 will include: paracetamol, ibuprofen, diclofenac. On stage 2: stage 1 + codeine and tramadol. On stage 3: stage 2 + morphine, fentanyl, oxycodone, pethidine. Oral and transcutaneous routes will be preferred to intravenous, intramuscular and subcutaneous. A need for elevation to the next step of analgesic ladder will be considered when the pain will be stronger than 6 points in Numeric Rating Scale (NRS) and will be present for more than 5 days.

INTERVENTIONS:
Procedure: Splanchnicectomy
  Arms: Surgical treatment

SUMMARY:
Pancreatic cancer is a difficult to treat disease, mainly due to the fact that diagnosis is made usually in the late stage of this condition. One of the treatment methods of pain accompanying this neoplasm is thoracoscopic splanchnicectomy. It has been shown that it is a safe procedure with a small percentage of complications, nevertheless it is often use as the last stage in pain management what significantly decreases its effectiveness.

The aim of this study is to determinate the effect of invasive pain treatment (splanchnicectomy) in patients with advanced pancreatic cancer on subjective pain perception at rest, in movement and after meals (measured with the BPI, QLQ- C30 and FACIT questionnaires), and suffering (measured with PRISM projection test), the use of painkillers during the disease and patients' overall survival. Moreover the investigators want to check if early performance of splanchnicectomy (on lower steps of analgesic ladder WHO) is combined with better therapeutic effect of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer
* Age over 18 years
* Signed informed consent to participate in the study

Exclusion Criteria:

* Age under 18 years
* Intellectual inability to fill the questionnaires
* Co-occurrence of a disease in which significant chronic pain exists, which was recognized before the onset of pancreatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-05 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain intensity at 1 year (BPI questionnaires) | one year

SECONDARY OUTCOMES:
Quality of life and pain intensity measurement (measured with the QLQ- C30, FACIT and BPI questionnaires) | From date of randomization until the date of death from any cause,assessed up to 100 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General, Endocrine and Transplant Surgery, Medical University of Gdansk., Gdansk, Poland

REFERENCES:
- [Derived] Dobosz L, Stefaniak T, Dobrzycka M, Wieczorek J, Franczak P, Ptaszynska D, Zasada K, Kanyion P. Invasive treatment of pain associated with pancreatic cancer on different levels of WHO analgesic ladder. BMC Surg. 2016 Apr 18;16:20. doi: 10.1186/s12893-016-0136-3. PMID 27090728